CLINICAL TRIAL: NCT04114903
Title: Exploring the Anti-inflammatory Properties of Cannabis and Their Relevance to Insulin Sensitivity
Acronym: SONIC
Status: Completed | Type: Observational
Sponsor: University of Colorado, Boulder (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Angela Bryan, PI, University of Colorado, Boulder
Other Study IDs: 1R01DA050515 (NIH)
Record Dates: First submitted 2019-09-06; First posted 2019-10-03 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes; Obesity; Cannabis Use; Insulin Sensitivity
Keywords: Diabetes; Obesity; Cannabis; Insulin Sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Insulin Resistance; Diabetes Mellitus; Marijuana Abuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples collected for insulin sensitivity, inflammation markers, and cannabinoid quantitation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study A: Adults balanced across the weight spectrum who have tried cannabis at least once with no negative reaction but are not regular users.
  Interventions: Other: Study A: Single use of cannabis flower product
- Study B: Sample of current cannabis users and non-users balanced across the weight spectrum who are matched on age, gender, BMI and physical activity.
  Interventions: Other: Study B: Ad libitum cannabis use for four weeks or no cannabis use

INTERVENTIONS:
Other: Study A: Single use of cannabis flower product — Participants are asked to purchase and use one of three cannabis flower strains with differing levels of THC and CBD: 1) CBD (~14% CBD/0% THC), 2) THC (~14% THC/0% CBD), or 3) THC+CBD (~7% THC/7% CBD).
  Groups: Study A
Other: Study B: Ad libitum cannabis use for four weeks or no cannabis use — Participants choose whether to use a cannabis flower product ad libitum for four weeks or to not use cannabis for four weeks. Participants who choose to use cannabis are asked to purchase and use one of three cannabis flower strains with differing levels of THC and CBD: 1) CBD (~14% CBD/0% THC), 2) THC (~14% THC/0% CBD), or 3) THC+CBD (~7% THC/7% CBD).
  Groups: Study B

SUMMARY:
This study tests the effects of cannabinoid levels in blood on inflammation and insulin sensitivity both acutely and chronically in individuals across the weight spectrum. To that end, the study employs two observational designs: 1) A study of acute effects with intermittent cannabis users and 2) A study in which current cannabis users will select one of three cannabis strains for four weeks and are compared to a matched control group who do not use cannabis to study chronic effects. Blood levels of THC and CBD, inflammatory biomarkers, and insulin resistance will be measured in both studies.

DETAILED DESCRIPTION:
According to the National Institute of Diabetes and Digestive and Kidney Diseases, over 30 million people in the US have diabetes, and just over 84 million people have pre-diabetes. Concurrently, 30 states and the District of Columbia have legalized cannabis for medical and/or recreational use and over the past decade, cannabis use among adults has more than doubled.

Public perception and some scientific data suggest that cannabis causes acute over-eating, creating concern that public and legal acceptance of cannabis use will worsen the obesity epidemic in the United States, where more than two-thirds of US adults (68.8%) are currently overweight or obese. Paradoxically, cross sectional data demonstrate associations between chronic cannabis use and lower body mass index (BMI), prevalence of obesity, insulin resistance, waist circumference, and actual rates of type 2 diabetes despite data supporting higher caloric intake acutely.

This study examines the effects of cannabinoid levels in blood on inflammation and insulin sensitivity both acutely and chronically in individuals across the weight spectrum. To that end, the study employs two observational designs: 1) A study of acute effects with intermittent cannabis users and 2) A study in which current cannabis users will select one of three cannabis strains for four weeks and are compared to a matched control group who do not use cannabis to study chronic effects.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Cannabis users in Study A must have smoked or vaped cannabis at least once since January 1st 2014 with no negative effects but NOT used in the past three months
* Cannabis users in Study B must have been a regular (at least weekly) user for at least a year
* Non-users in Study B cannot have used any cannabis in the previous year
* Weight stable (<5 pound fluctuation in the past six months)
* Planning to remain in the Boulder-Denver area for the next month
* Fasting blood glucose greater than or equal to 55 mg/dl and less than or equal to 126 mg/dl
* Cannabis users in Study A must endorse knowledge of the procedure(s) for smoking or vaping cannabis

Exclusion Criteria:

* Known auto-immune disease
* Report of other drug use (cocaine, opiates, methamphetamine) in the past 90 days or fail urine screen for any of these drugs
* Daily tobacco (cigarette, E-cigs, smokeless) user, given the impact of tobacco smoking on insulin function
* Blood alcohol level greater than 0 at screening
* Current use of medications for glucose lowering, immunosuppression, or anti-inflammation
* Acute illness
* Current use of psychotropic medications
* Current diagnosis of diabetes
* Heavy drinking as defined by an Alcohol Use Disorders Test (AUDIT)
* Females can not be pregnant or trying to become pregnant
* Females can not be nursing mothers
* Have donated blood in the 8 weeks before the study or intend to donate blood in the 8 weeks after the study.

Ages: 21 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Markers of Inflammation | Study A: Difference between cytokines at baseline and cytokines one week later after acute use of cannabis product. Study B: Change from baseline to four weeks
  Change in Circulating Levels of Cytokines (TNF-α, IL-1B, IL-4, IL-6, IL-10, IL-13, MCP-1)
Change in Matsuda Index of Insulin Sensitivity | Study A: Baseline versus after acute use one week later of cannabis product. Study B: The two tests will be separated by four weeks
  Calculation of Insulin Sensitivity using changes in fasting plasma glucose (FPG) and fasting plasma insulin (FPI).
  Measurements are collected on venous blood samples at 0, 30, 60, 90, and 120 minutes after ingestion of 75 grams oral glucose during oral glucose tolerance test (OGTT)
  Matsuda Index is calculated as follows: 10000/sqrt ((FPG X FPI) X (Mean OGTT glucose concentration X Mean OGTT insulin concentration))
Change in Plasma Glucose | Study A: Baseline versus one week later after acute use of cannabis product. Study B: The two tests will be separated by four weeks
  Change in glucose over time after ingestion of 75 grams oral glucose measured during during oral glucose tolerance test (OGTT). Measurements are collected on venous blood samples at 0, 30, 60, 90, and 120 minutes.
Change in Plasma Insulin | Study A: Baseline versus one week later after acute use of cannabis product. Study B: The two tests will be separated by four weeks
  Change in insulin over time after ingestion of 75 grams oral glucose measured during OGTT. Measurements are collected on venous blood samples at 0, 30, 60, 90, and 120 minutes.

SECONDARY OUTCOMES:
Stanford Seven-Day Physical Activity Recall (PAR) | Study A: Baseline and one week following baseline Study B: Baseline and four weeks following baseline
  Interviewer administered assessment of number of minutes of mild, moderate, and vigorous physical activity over the previous seven days.
Sleep Quality | Study A: Baseline to one week following baseline Study B: Baseline to four weeks following baseline
  Pittsburgh Sleep Quality Index: Measurement of the quality and patterns of sleep from poor to good measuring seven domains (e.g., latency, duration, disturbances) over the last 2 weeks.
Marijuana Consumption Questionnaire | Study A: Baseline and one week following baseline Study B: Baseline and four weeks following baseline
  Frequency and quantity of cannabis use, age of first use, peer use, perceived risk from cannabis, and perceived availability of cannabis
Marijuana Dependence Scale | Study A: Baseline and one week following baseline Study B: Baseline and four weeks following baseline
  Based on DSM V criteria that were converted to a self-report to assess dependence and other problems related to the use of cannabis
Marijuana Withdrawal Checklist | Study A: Baseline and one week following baseline Study B: Baseline and four weeks following baseline
  A 15-item scale used to collect information on withdrawal symptoms participants may be experiencing due to lack of use of marijuana
The Alcohol Use Disorder Identification Test (AUDIT) | Study A: Baseline and one week following baseline Study B: Baseline and four weeks following baseline
  Standardized assessment of the extent of alcohol use and problems related to alcohol use
Timeline Follow-Back of Substance Use | Study A: Baseline and one week following baseline Study B: Baseline and four weeks following baseline
  Calendar-based assessment of daily substance use for the 30 days prior to the baseline session only for both studies
SF-12 Health Survey | Study A: Baseline and one week following baseline Study B: Baseline and four weeks following baseline
  The SF-12 Health Survey is a 12-item questionnaire used to assess general health and well-being and includes domains of physical functioning, role-physical, pain, general health, vitality, social functioning, role-emotional and mental health
Nutrition Data System for Research 24-Hour Dietary Recall | Study A: Baseline and one week following baseline Study B: Baseline and four weeks following baseline
  Interviewer administered recall measure developed by the University of Minnesota Nutrition Coordinating Center (NCC), that facilitates the standardized collection of 24-hour dietary recall data
Stanford Leisure-Time Activity Categorical Item (L-Cat) | Study A: Baseline and one week following baseline Study B: Baseline and four weeks following baseline
  Self-report measure of a single item comprising six descriptive categories ranging from inactive to very active

OTHER OUTCOMES:
Daily online survey of cannabis use, alcohol use, exercise and diet | Study B only: Daily for four weeks between baseline and second study visit
  Daily surveys sent to Study B participants during the four-week period between study visits querying for cannabis use, alcohol use, minutes of exercise, and consumption of fruits and vegetables

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Innovation and Creativity, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No